CLINICAL TRIAL: NCT05569629
Title: Diagnostic Yield of Bronchial Washing Before and After Endobronchial Biopsy and Bronchial Brushing for Endoscopically Visible Tumours
Brief Title: Bronchial Washing Beforeand After Endobronchial Biopsy and Bronchial Brushing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Clinical Lecturer, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: PrePostBW
Record Dates: First submitted 2022-10-02; First posted 2022-10-06 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Toothbrushing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All bronchial washing samples will be examined independently by two senior pathologists, who will be blinded to the sequence of bronchial washing and results of the other samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre & post-EBBx/BB group (Experimental): BW will be performed once before endobronchial biopsy and bronchial brushing, and once after endobronchial biopsy and bronchial brushing
  Interventions: Procedure: Bronchial washing before endobronchial biopsy and brushing
- Post-EBBx/BB group (No Intervention): BW will be performed once after endobronchial biopsy and bronchial brushing

INTERVENTIONS:
Procedure: Bronchial washing before endobronchial biopsy and brushing — Bronchial washing: adding bronchial washing once to the standard endoscopic sampling sequence (endobronchial biopsy and brushing first, followed by bronchial washing once) in the experimental arm
  Arms: Pre & post-EBBx/BB group

SUMMARY:
Objective: To identify the optimal position of bronchial washing (BW) in the sequence of bronchoscopic sampling in order to maximize the ability to confirm malignancy for endoscopically visible tumours.

Hypothesis to be tested: The investigators hypothesize that the diagnostic yield, with the incorporation of contemporary cytology processing techniques, of combined BW before and after endobronchial biopsy (EBBx) / bronchial brushing (BB) is higher than that of single BW after EBBx / BB.

Design and subjects: This is a prospective, randomized controlled study to be conducted in the medical department of a tertiary care hospital in Hong Kong involving patients who will receive bronchoscopy. Patients will be recruited if an endoscopically visible tumour is suspected.

Study instruments: Patients will be randomized into two groups. The diagnostic yield of confirming malignancy for endoscopically visible tumours, with the incorporation of contemporary cytology processing techniques, will be compared between obtaining BW before and after EBBx / BB, and obtaining single BW after EBBx / BB.

Main outcome measures: Only patients with a definite cytological or histological diagnosis of lung cancer will be included in further analyses. The diagnostic yield of diagnosing lung cancer between the pre & post-EBBx/BB group and post-EBBx/BB group will be compared by the Chi-square test as an intergroup comparison.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer in Hong Kong, and also ranks first in cancer-related mortality. Early diagnosis of lung cancer is pivotal to facilitating early treatment and ensuring a better prognosis. In those centrally located tumours, especially those arising from the bronchus and endoscopically visible, bronchoscopy with endobronchial biopsy (EBBx), bronchial brushing (BB) and bronchial washing (BW) are the three major endoscopic techniques to establish the pathological diagnosis. The diagnostic yield of EBBx is the highest among the three, ranging from 48% to 79%, but occasionally fails to give the proper diagnosis because of thick necrotic materials covering the tumours, crushed artefacts and inappropriate targeting. Supplementing BW, a cost-effective procedure, can increase the overall diagnostic yield by 2% to 12% beyond EBBx alone. The final diagnostic yield can be as high as up to 97% for endoscopically visible tumours by combining EBBx, BB and BW in a single bronchoscopy procedure. Therefore, various guidelines recommend performing these three procedures to maximize the diagnostic yield and the volume of tissue obtained for phenotyping and genotyping of advanced non-small cell lung carcinoma.

The sequence of these three endoscopic sampling techniques, especially the relative position of BW, has been controversial. BW obtains the return of normal saline after instilling over an endoscopically visible tumour, which contains exfoliated malignant cells from the tumour. It is logical that the shedding of malignant cells is increased after breaking or ablating the bronchial mucosa by EBBx and BB (EBBx / BB), but this hypothesis was not supported by several prospective studies. However, these studies were limited by inconsistent incorporation of BB, and a majority of them were self-controlled comparative studies. The only randomized, multi-centre study by Lee et al showed no significant difference in the diagnostic yield of BB before and after EBBx, but again, BB was not consistently performed in the study. Instead, the diagnostic yield by combining the BW before and after EBBx, with or without BB, was higher than a single BW alone. Although the BW obtained after EBBx / BB was more haemorrhagic in appearance, the interpretation was considered unaffected. Guidelines for bronchoscopy addressing the sequence of endoscopic sampling are conflicting. BTS guideline commented that the sequence of sample acquisition is not important, while the Indian guideline recommends BW should be performed both before and after EBBx / BB. The guideline issued by the American College of Chest Physicians did not address this issue. Nowadays, more sophisticated endoscopic sampling techniques, e.g. cryobiopsy, are available with a high diagnostic yield, but they usually carry higher procedural risk and are only available in tertiary centres with expertise. Therefore, it is necessary to optimize the sampling sequence with existing and widely available techniques.

The method of cytological processing plays a critical part in optimizing the diagnostic yield of BW. Conventional cytology (CC) preparation was employed in the above-mentioned studies, and the authors did not address the reason for negative BW cytology. Only Van der MA drift et al identified the problem of poor cellularity in a number of negative BW specimens. In the past decade, the introduction of liquid-based cytology (LBC) and cell block (CB) preparation to reduce unsatisfactory cytological results and eliminate obscuring factors such as blood, inflammation, and mucus has improved the overall diagnostic yield in addition to CC. CB also serves as another source of diagnostic material for immunohistochemical (IHC) and molecular studies. The recent developments in whole-slide scanners with increased throughput and z-stacking three-dimensionally reconstructed images allow for accurate and reproducible cellular quantification and cytomorphometric analysis. Digital pathology-based quantification can complement, validate and provide added analysis to the yield, diagnostic accuracy and cytological effects in different protocols for bronchoscopic sampling. With the incorporation of LBC and CB techniques and an optimal sequence of bronchoscopic sampling, the diagnostic accuracy, cellular yield and specimen quality can be further improved and guide personalized oncological treatment.

The investigators believe that combining EBBx and BB together is important to ablate a larger area of bronchial mucosa than either procedure alone, and potentially release more malignant cells during the BW. To date, there is no randomized controlled trial comparing the diagnostic yield of combined BW before and after EBBx / BB, and BW after EEBx / BB. The investigators hypothesize that the diagnostic yield, with the incorporation of contemporary cytology processing techniques, of combined BW before and after EBBx / BB is higher than that of single BW after EBBx / BB. The aim of this study is to identify the optimal position of BW in the sequence of bronchoscopic sampling in order to maximize the ability to confirm malignancy for endoscopically visible tumours.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for bronchoscopy and endoscopic sampling procedures (i.e. endobronchial biopsy (EBBx), bronchial brushing (BB) and bronchial washing (BW)) as recommended by the prevailing local guideline
* Patients will undergo endoscopic sampling procedures to the airway that contains the endoscopically visible tumours
* Patients who are aged 18 years old or above
* Patients are cognitively capable to consent for the procedure and the study
* Patients with endoscopically visible tumours in the airway during bronchoscopy, that can be approached by endoscopic sampling procedures
* Only those visible lesions with endoscopic morphology of tumorous, infiltrative, necrotic-coated types will be included

Exclusion Criteria:

* Endoscopically visible tumours are not expected based on pre-bronchoscopy imaging (e.g. CT thorax)
* Failed to obtain informed consent due to patient's refusal or cognitive impairment
* Bronchoscopy that will be performed in an emergency situation that precludes a detailed examination or prolonged procedure time, e.g. massive haemoptysis
* The prevailing contraindications for bronchoscopy or bronchoscopic samplings, e.g. uncorrected coagulopathy, and uncontrolled respiratory failure
* Lesions with an anticipated high risk of severe bleeding are found, e.g. carcinoid tumour, Dieulafoy's lesion and Kaposi sarcoma
* The targeted lesion is located in the trachea or carina
* Patients with tumours morphology of submucosal type or extrinsic compressions, or with a normal mucosal appearance in the targeted airway
* Technical reasons precluding an optimal sampling of the lesion by endoscopic sampling procedures, including sharp angulation of the airway and patient intolerance
* Excessive bleeding due to EBBx and BB causing difficult procedure of subsequent BW or premature termination of the procedure
* Coexisting tumours in the same lobar or segmental bronchi, either proximal or distal to the targeted lesion, as it is impossible to distinguish the source of exfoliated cells
* A total volume of more than 100mL of normal saline is instilled for the first BW in the combined BW group, as the total amount of normal saline after the two BW procedures may exceed 200mL and impose a risk of impaired gaseous exchange

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
To compare the diagnostic yield of bronchial washing in confirming malignancy (intergroup comparison) | 18 months
  To compare the diagnostic yield of bronchial washing in confirming malignancy for endoscopically visible tumours between obtaining bronchial washing before and after endobronchial biopsy and bronchal brushing, and obtaining single bronchial washing after endobronchial biopsy and bronchal brushing

SECONDARY OUTCOMES:
To compare the diagnostic yield of bronchial washing in confirming malignancy (intragroup comparison) | 18 months
  To compare the diagnostic yield of bronchial washing in confirming malignancy for endoscopically visible tumours between obtaining bronchial washing once before endobronchial biopsy and bronchal brushing and obtaining single bronchial washing after endobronchial biopsy and bronchal brushing
To compare the cell adequacy in the bronchial washing cytology specimens | 18 months
  To compare the cell adequacy in the bronchial washing cytology specimens obtained before and after endobronchial biopsy and bronchal brushing, and obtaining single bronchial washing after endobronchial biopsy and bronchal brushing
To compare the time spent for endoscopic sampling procedures | 18 months
  To compare the time spent for endoscopic sampling procedures between obtaining the bronchial washing cytology specimens before and after endobronchial biopsy and bronchal brushing, and obtaining single bronchial washing after endobronchial biopsy and bronchal brushing
To compare the occurrence of bleeding complications during endoscopic sampling procedures | 18 months
  To compare the occurrence of bleeding complications during endoscopic sampling procedures between obtaining the bronchial washing cytology specimens before and after endobronchial biopsy and bronchal brushing, and obtaining single bronchial washing after endobronchial biopsy and bronchal brushing

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Study Director — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No